CLINICAL TRIAL: NCT05863273
Title: Real World Study on the Efficacy and Safety of Apremilast in Chinese Patients With Moderate to Severe Plaque Psoriasis, a Multi Center, Prospective, Observational Trial（REACT）
Status: Completed | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Collaborators: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Xing hua Gao, First Hospital of China Medical University, First Hospital of China Medical University
Other Study IDs: OTL-A-2201
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis
Keywords: Apremilast; Otazla; Real World Study
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Apremilast: Dosage of Apremilast（Otezla®） from 10mg qd, titrate to recommended dosage of 30 mg BID，recommended by specification.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Dosage of Apremilast（Otezla®） from 10mg qd, titrate to recommended dosage of 30 mg BID，recommended by specification.

SUMMARY:
This is a multicenter, one-arm, prospective, observational study，intended to assess evaluation of efficacy and safety of Apremilast in Chinese patients with moderate-to-severe plaque psoriasis。During this study, it is expected to collect data at at baseline and weeks 2, 6, 10, 16, and 20 after treatment。

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ≥ 18 years of age at the time of signing the informed consent document；
* Patients with moderate-to-severe plaque psoriasis：Simultaneously meet (1)and (2): (1)PASI≥ 3；(2) DLQI ≥ 6；
* Subject is a candidate for phototherapy and/or systemic therapy
* Patients who wish to be treated with Apremilast and sign the informed consent

Exclusion Criteria:

* Allergy to Apremilast or any component of the study drug；
* Use of phototherapy within 4 weeks prior to randomization；Use of systemic drugs or biologic agents within 4 half-life periods prior to randomization；Patients with inadequate response or intolerance to previous systemic therapy do not need to consider drug washout；
* Currently using potent cytochrome P450 enzyme inducers (e.g., rifampin, phenobarbital, carbamazepine, phenytoin, etc.)；
* History of substance abuse, suicide attempts, or mental illness；
* Patients who are currently pregnant, breastfeeding, or planning a pregnancy during the study observation period；
* Pustular type, erythroderma type and other psoriasis patients；
* Other circumstances that investigators don't consider appropriate to include.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with moderate to severe plaque psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
DLQI or PASI improvement | 16 week
  At week 16，Proportion of patients with DLQI improvement (DLQI ≤5 or DLQI improvement by ≥4 points from baseline) or PASI improvement (PASI <3)

SECONDARY OUTCOMES:
PASI, PGA, BSA, DLQI, pruritus VAS and pain VAS | 16 week
  Absolute values of change from baseline in PASI, PGA, BSA, DLQI, pruritus VAS and pain VAS in subjects at week 16 of treatment
DLQI improvement | 2 week
  Proportion of patients with DLQI score ≤5 or improvement ≥4 points from baseline at each visits
DLQI improvement | 6 week
  Proportion of patients with DLQI score ≤5 or improvement ≥4 points from baseline at each visits
DLQI improvement | 10 week
  Proportion of patients with DLQI score ≤5 or improvement ≥4 points from baseline at each visits

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Gao, MD, Study Director — First Hospital of China Medical University
Locations (2):
- China (2):
  - the First Hospital of China Medical University, Shenyang, China
  - China-Japan Friendship Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No